CLINICAL TRIAL: NCT02540798
Title: Do Increased Levels of Anxiety Decrease the Reproducibility of Symptoms During Urodynamic Studies in Women?
Brief Title: Do Patient Anxiety Levels Decrease Urodynamic Test Reproducibility?
Status: Completed | Type: Observational
Sponsor: Sandwell & West Birmingham Hospitals NHS Trust (Other)
Collaborators: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Stephanie Smith, Trainee Clinical Scientist, Sandwell & West Birmingham Hospitals NHS Trust
Other Study IDs: SandwellWBNHS
Record Dates: First submitted 2015-08-07; First posted 2015-09-04 (Estimated); Last update posted 2016-10-24 (Estimated); Status verified 2016-10

CONDITIONS: Anxiety; Overactive Bladder; Urinary Incontinence, Stress; Urinary Incontinence, Urge; Urinary Retention
Keywords: Anxiety; Urodynamics; Symptom reproducibility; Lower urinary tract symptoms; Women
MeSH Terms: conditions — Anxiety Disorders; Urinary Bladder, Overactive; Urinary Incontinence, Stress; Urinary Incontinence, Urge; Urinary Retention; Lower Urinary Tract Symptoms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
This study will look at how pre-test anxiety levels affect the reproducibility of symptoms during routine urodynamic testing in women. Urodynamics is a test that assesses the function of the lower urinary tract, including the bladder.

DETAILED DESCRIPTION:
The results of urodynamic tests often determine treatment for patients, which may include bladder retraining, medication and/or surgery. Thus, it is important for the results of urodynamics to be accurate and representative of the patient's symptoms outside of the clinic.

Pre-test anxiety levels in women undergoing urodynamics will be measured using a validated questionnaire HADS (Hospital anxiety and depression scale). The patient, prior to their routine urodynamics test, will fill out this self-administered questionnaire.

Reproducibility of patient symptoms will be measured using a non-validated quantitative bladder test assessment. The patient will fill out this self-administered quantitative bladder assessment after their urodynamics test.

The pre-test anxiety and symptom reproducibility variables will be correlated against each other to assess whether there is correlation between the two. A Spearman Rho test will be used to assess the strength of the relationship.

ELIGIBILITY:
Inclusion Criteria:

* Women attending for their first time to the urodynamics clinic for the assessment of their bladder function
* Must be over the age of 18 years old
* Must be able to consent for themselves

Exclusion Criteria:

* Any patients not covered in the inclusion criteria

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Only patients referred for urodynamics for the first time will be asked to consider being included in the study. Minimum of 30 participants to be included. Recruited via obstetric and urogynaecology clinics.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2015-07; Primary Completion 2015-11 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Correlate pre-test anxiety scores with the reproducibility of symptom scores from urodynamic studies in women | 9 months

SECONDARY OUTCOMES:
The number of women who have their typical symptoms reproduced during urodynamic studies | 9 months
Number of women with abnormal (i.e. not normal) urodynamic diagnosis and high pre-test anxiety scores | 9 months
Number of women with abnormal (i.e. not normal) urodynamic diagnosis with low reproducibility of symptom scores | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Victor Olagundoye, Principal Investigator — Sandwell and West Birmingham Hospitals NHS Trust
Locations (1):
- Sandwell and West Birmingham Hospitals NHS Trust, Birmingham, United Kingdom